CLINICAL TRIAL: NCT06686888
Title: The Impact of Short-Chain Fatty Acids on the Gut Hormone Release After Delivery in the Small Intestine and Colon
Brief Title: The Impact of Short-Chain Fatty Acids on Gut Hormone Release After Delivery in the Small and Large Intestine of Healthy Volunteers
Acronym: Histine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S67256- study 2
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Satiety Hormones; Short-chain Fatty Acids; Satiety and Appetite; Intestinal Absorption; Metabolism; Glucose Homeostasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Small intestinal delivery capsules (Experimental): SCFA
  Interventions: Dietary Supplement: SCFA
- Colon-delivery capsules (Experimental): SCFA
  Interventions: Dietary Supplement: SCFA
- placebo capsules (Placebo Comparator): Microcristalline cellulose
  Interventions: Dietary Supplement: microcristalline cellulose

INTERVENTIONS:
Dietary Supplement: SCFA — On test days participants will ingest the capsules during a standard no fiber breakfast. Blood samples will be collected at regular time points for 8 hours. A visual analogue scale that questions hunger and satiety will be completed at regular time points.
  Arms: Colon-delivery capsules; Small intestinal delivery capsules
Dietary Supplement: microcristalline cellulose — On test days participants will ingest the capsules during a standard no fiber breakfast. Blood samples will be collected at regular time points for 8 hours. A visual analogue scale that questions hunger and satiety will be completed at regular time points.
  Arms: placebo capsules

SUMMARY:
The goal of this crossover study is to evaluate the impact of short-chain fatty acids (SCFA) on the gut hormone release after administration in the small intestine or colon in healthy participants. The main question it aims to answer is whether the site of administration of SCFA affects the gut hormone release. On test days participants will ingest capsules filled with SCFA that are specifically delivered in the small intestine or the colon. Subsequently, blood samples are collected at regular time points.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* healthy
* normal BMI (18.5-25 kg/m^2)
* age within 18-50 years

Exclusion Criteria:

* Chronic gastrointestinal disorders such as inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), celiac disease, chronic constipation (less than 3 stools a week) and chronic frequent diarrhoea (more than 3 stools a day)
* Previous abdominal surgery, except from appendectomy
* Being on a weight loss, gluten-free, lactose-free, or vegan diet
* The donation of blood during the last 3 months or suffering from low blood haemoglobin levels
* The use of antibiotics or other medication that affects the gastrointestinal tract 3 months preceding the study and/or during the study
* The use of prebiotics or probiotics 2 weeks preceding the study and/or during the study
* Pregnancy, lactation or wish to become pregnant during the study period
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The release of gut hormones | 8 hours
  Gut hormone GLP-1 (pmol/l) and PYY (pg/ml) concentrations will be quantified in the blood samples collected at different time points.

SECONDARY OUTCOMES:
The glycemic and insulinemic response | 8 hours
  The glucose (mg/dl) and c-peptide (nmol/l) concentration will be determined in blood samples collected at regular time points during the test day

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.